CLINICAL TRIAL: NCT00602459
Title: A Genetic Risk-Stratified, Randomized Phase II Study of Four Fludarabine/Antibody Combinations for Patients With Symptomatic, Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Fludarabine and Rituximab With or Without Lenalidomide or Cyclophosphamide in Treating Patients With Symptomatic Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00441; NCI-2009-00441 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000584205; ECOG-10404; SWOG-C10404; 11-00126; SWOG C10404; ECOG 10404; CAN-NCIC-CL3; CALGB 10404 (Other: Alliance for Clinical Trials in Oncology); CALGB-10404 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine phosphate; Lenalidomide; Rituximab; CT-P10

ARMS (4):
- Arm A (rituximab, fludarabine phosphate) (Active Comparator): Participants receive induction therapy (every 28 days for up to 6 cycles) of: Patients receive rituximab IV over 1-4 hours on days 1 (50 mg/m^2), 3 (325 mg/m^2), and 5 (375 mg/m^2) of course 1 and on day 1 (375 mg/m^2) of all subsequent courses. Patients also receive fludarabine phosphate 25 mg/m^2/day IV over 30 minutes or PO on days 1-5.
  Interventions: Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Rituximab
- Arm B (rituximab, fludarabine phosphate, lenalidomide) (Experimental): Participants receive induction therapy (every 28 days for up to 6 cycles) of: rituximab IV over 1-4 hours on days 1 (50 mg/m^2), 3 (325 mg/m^2), and 5 (375 mg/m^2) of course 1 and on day 1 (375 mg/m^2) of all subsequent courses. Patients also receive fludarabine phosphate 25 mg/m^2/day IV over 30 minutes or PO on days 1-5. Participants without progression receive consolidation therapy lenalidomide 5mg/day cycle 1, 10 mg/day cycles 2-6 PO QD on days 1-21 of 28 day cycle.
  Interventions: Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Rituximab
- Arm C (rituximab, fludarabine phosphate, cyclophosphamide) (Experimental): Participants receive induction therapy (every 28 days for up to 6 cycles) of: rituximab IV over 4 hours on days 1 (50mg/m^2) and 3 (325 mg/m^2) of course 1 and on day 1 (500 mg/m^2) of all subsequent courses. Patients then receive fludarabine phosphate (age < 70: 25 mg/m^2/day; age >= 70: 20 mg/m^2/day) IV piggyback over 30 minutes or PO (32 mg/m^2/day) followed by cyclophosphamide (age < 70: 250 mg/m^2/day; age >= 70: 150 mg/m^2/day) IV piggyback over 30 minutes on days 1-3.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Rituximab
- Arm D (rituximab, fludarabine, cyclophosphamide, lenalidomide) (Experimental): Patients receive the first course of induction therapy as in Arm A or B before being re-assigned to Arm D. Beginning in course 2, patients receive rituximab IV (500 mg/m^2) on day 1 and fludarabine phosphate (age < 70: 25 mg/m^2/day; age >= 70: 20 mg/m^2/day) IV piggyback over 30 minutes or PO (32 mg/m^2/day) and cyclophosphamide IV (age < 70: 250 mg/m^2/day; age >= 70: 150 mg/m^2/day) piggyback over 30 minutes on days 1-3. Participants without progression receive consolidation therapy: lenalidomide 5mg/day cycle 1, 10 mg/day cycles 2-6PO QD on days 1-21 of 28 day cycle.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm C (rituximab, fludarabine phosphate, cyclophosphamide); Arm D (rituximab, fludarabine, cyclophosphamide, lenalidomide)
Drug: Fludarabine Phosphate — Given IV or PO
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm B (rituximab, fludarabine phosphate, lenalidomide); Arm D (rituximab, fludarabine, cyclophosphamide, lenalidomide)
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima

SUMMARY:
This randomized phase II trial studies how well fludarabine (fludarabine phosphate) and rituximab with or without lenalidomide or cyclophosphamide work in treating patients with symptomatic chronic lymphocytic leukemia. Drugs used in chemotherapy, such as fludarabine phosphate and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. Giving fludarabine phosphate and rituximab together with lenalidomide or cyclophosphamide may be an effective treatment for chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the two-year progression-free survival (PFS) after remission induction with four different chemo-immunotherapy combinations for patients with untreated, symptomatic, lower-risk and high-risk chronic lymphocytic leukemia (CLL) to decide which of the four arms, if any, to take forward into a randomized phase III trial.

II. To determine the induction response to fludarabine phosphate and rituximab (FR) and fludarabine phosphate, cyclophosphamide, and rituximab (FCR) in each of these arms, along with the consolidation response to lenalidomide in patients with CLL.

III. To determine the toxicity from these four chemoimmunotherapy combinations and that of consolidation therapy with lenalidomide.

IV. To determine the induction response and toxicity of FCR in patients with deletion (del) (11q22.3) along with consolidation response, 2-year PFS and toxicity of lenalidomide in this specific genetic group.

V. To determine the effect of pretreatment biologic characteristics on clinical outcomes, such as attaining a complete response to induction therapy and progression-free survival.

VI. To collect relapse samples to determine the frequency of clonal evolution among patients with immunoglobulin heavy chain variable region (IgVH) mutated and unmutated disease and to study mechanisms of resistance to chemoimmunotherapy.

VII. To determine if flow cytometry-negative status immediately post-therapy and at 24 months after study entry is an effective surrogate marker for prolonged progression-free survival and overall survival.

OUTLINE: Patients are randomized to 1 of 3 treatment arms (Arms A, B, or C). Patients on Arm A or B who are found to be del (11q22.3) positive are assigned to Arm D beginning with course 2 of induction therapy.

ARM A (remission-induction [RI] therapy with fludarabine phosphate and rituximab): Participants receive induction therapy (every 28 days for up to 6 cycles) of: rituximab intravenously (IV) over 1-4 hours on days 1 (50 mg/m^2), 3 (325 mg/m^2), and 5 (375 mg/m^2) of course 1 and on day 1 (375 mg/m^2) of all subsequent courses. Patients also receive fludarabine phosphate 25 mg/m^2/day IV over 30 minutes or orally (PO) on days 1-5.

ARM B (RI therapy with fludarabine phosphate and rituximab followed by remission-consolidation [RC] therapy with lenalidomide): Participants receive induction therapy (every 28 days for up to 6 cycles) of: rituximab IV over 1-4 hours on days 1 (50 mg/m^2), 3 (325 mg/m^2), and 5 (375 mg/m^2) of course 1 and on day 1 (375 mg/m^2) of all subsequent courses. Patients also receive fludarabine phosphate 25 mg/m^2/day IV over 30 minutes or PO on days 1-5. Participants without progression receive consolidation therapy: lenalidomide 5mg/day cycle 1, 10 mg/day cycles 2-6 PO once daily (QD) on days 1-21 of 28 day cycle.

ARM C (RI therapy with fludarabine phosphate, rituximab, and cyclophosphamide): Participants receive induction therapy (every 28 days for up to 6 cycles) of: rituximab IV over 4 hours on days 1 (50mg/m^2) and 3 (325 mg/m^2) of course 1 and on day 1 (500 mg/m^2) of all subsequent courses. Patients then receive fludarabine phosphate (age < 70: 25 mg/m^2/day; age >= 70: 20 mg/m^2/day) IV piggyback over 30 minutes or PO (32 mg/m^2/day) followed by cyclophosphamide (age < 70: 250 mg/m^2/day; age >= 70: 150 mg/m^2/day) IV piggyback over 30 minutes on days 1-3.

ARM D (RI therapy with fludarabine phosphate, rituximab, and cyclophosphamide followed by RC therapy with lenalidomide): Patients receive the first course of induction therapy as in Arm A or B before being re-assigned to Arm D. Beginning in course 2, patients receive rituximab IV (500 mg/m^2) on day 1 and fludarabine phosphate (age < 70: 25 mg/m^2/day; age >= 70: 20 mg/m^2/day) IV piggyback over 30 minutes or PO (32 mg/m^2/day) and cyclophosphamide IV (age < 70: 250 mg/m^2/day; age >= 70: 150 mg/m^2/day) piggyback over 30 minutes on days 1-3. Participants without progression receive consolidation therapy: lenalidomide 5mg/day cycle 1, 10 mg/day cycles 2-6 PO QD on days 1-21 of 28 day cycle.

After completion of study therapy, patients are followed up every 3 months for 1 year and then every 6 months for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Specific diagnosis of B-cell CLL:

  * An absolute lymphocytosis of > 5,000/uL

    * Morphologically, the lymphocytes must appear mature with < 55% prolymphocytes
    * Bone marrow examination must include at least a unilateral aspirate and biopsy; the aspirate smear must show > 30% of all nucleated cells to be lymphoid or the bone marrow core biopsy must show lymphoid infiltrates compatible with marrow involvement by CLL; overall cellularity must be normocellular or hypercellular
    * Local institution lymphocyte phenotype must reveal a predominant B-cell monoclonal population sharing a B-cell marker (cluster of differentiation [CD]19, CD20, CD23) with the CD5 antigen, in the absence of other pan-T-cell markers; additionally, the B-cells must be monoclonal with regard to expression of either kappa or lambda and have surface immunoglobulin expression of low density; patients with bright surface immunoglobulin levels must have CD23 co-expression
* Patients must have symptomatic and active intermediate or high-risk categories of the modified three-stage Rai staging system:

  * Not eligible: low risk, Rai stage 0, lymphocytes (L) in blood (> 5000/uL) and marrow (> 30%) only
  * Intermediate risk, Rai stage I, L + enlarged lymph nodes (LN)
  * Intermediate risk, Rai stage II, L + spleen and/or liver (LN + or -)
  * High risk, Rai stage III, L + anemia (hemoglobin < 11 gm/dL)
  * High risk, Rai stage IV, L + thrombocytopenia (platelets < 100,000/uL)
* Patients in the intermediate-risk group must have evidence of active disease as demonstrated by at least one of the following criteria:

  * Massive or progressive splenomegaly, hepatomegaly and/or lymphadenopathy
  * Presence of weight loss > 10% over the preceding 6 month period
  * Grade 2 or 3 fatigue
  * Fevers > 100.5 degrees Fahrenheit (°F) or night sweats for greater than 2 weeks without evidence of infection
  * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of less than 6 months
* No prior therapy for CLL, including no corticosteroids for autoimmune complications that have developed since the initial diagnosis of CLL
* No medical condition requiring chronic use of oral corticosteroids
* Performance status 0 - 2
* Patients with human immunodeficiency virus (HIV) infection may be eligible provided they meet the following criteria: no evidence of infection with hepatitis B or C; CD4+ cell count > 350/mm^3; no evidence of resistant strains of HIV; if not on anti-HIV therapy, an HIV viral load < 10,000 copies HIV ribonucleic acid (RNA)/mL; if on HIV therapy, HIV viral load < 50 copies HIV RNA/mL; and no history of acquired immune deficiency syndrome (AIDS)-defining condition; patients receiving concurrent zidovudine or stavudine may not be enrolled
* Non-pregnant and non-nursing
* In females of child-bearing potential randomized to Arm B or assigned to Arm D, a negative urine or serum pregnancy test with a sensitivity of at least 25 mIU/mL will be required: 1) 10-14 days prior to beginning lenalidomide consolidation therapy; and 2) within 24 hours prior to the first dose of lenalidomide consolidation therapy; in addition, females of childbearing potential in Arm B and Arm D with regular menses must have a pregnancy test performed weekly during the first 28 days of treatment, and then every 28 days while taking lenalidomide (including breaks in lenalidomide), at discontinuation of lenalidomide, and then 28 days following discontinuation of lenalidomide; if menses are irregular, a pregnancy test must be performed weekly during the first 28 days of treatment, and then every 14 days while taking lenalidomide, at discontinuation of lenalidomide, and at 14 and 28 days after discontinuation of lenalidomide; additionally, females of childbearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO reliable methods of birth control - one highly effective method (intrauterine device [IUD], hormonal [birth control pills, injections, or implants], tubal ligation, or partner's vasectomy), and one additional effective method (latex condom, diaphragm, or cervical cap) - AT THE SAME TIME, at least 4 weeks before she begins lenalidomide therapy, while participating in the study, and for at least 4 weeks after completing lenalidomide therapy; "females of childbearing potential" is defined as a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy, or who has had menses at any time in the preceding 24 consecutive months (not been naturally postmenopausal for at least 24 consecutive months)
* Male patients randomized to Arm B or reassigned to Arm D must agree not to father a child and to use a latex condom during any sexual contact with females of childbearing potential while taking lenalidomide and for at least 4 weeks following completion of lenalidomide therapy, even if the patient have undergone a successful vasectomy
* All patients randomized to Arm B or reassigned to Arm D must be counseled by a trained counselor every 28 days during consolidation therapy about pregnancy precautions and risks of fetal exposure
* Creatinine =< 1.5 x upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2008-01-15 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Byrd, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (364):
- United States (355):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Unspecified Site, Rockville, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - McGill University Health Centre at Royal Victoria Hospital, Montreal, Quebec
  - CHU de Quebec-Hopital du Saint-Sacrement (HSS), Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2008 to August 2012, 418 participants were recruited to this study.
Groups:
- Arm A (Rituximab, Fludarabine Phosphate): Participants receive induction therapy (every 28 days for up to 6 cycles) of: rituximab IV over 1-4 hours on days 1 (50 mg/m^2), 3 (325 mg/m^2), and 5 (375 mg/m^2) of course 1 and on day 1 (375 mg/m^2) of all subsequent courses. Patients also receive fludarabine phosphate 25 mg/m^2/day IV over 30 minutes or PO on days 1-5.
Period: Initial Registration/Randomization
Arm/Group | Arm A (Rituximab, Fludarabine Phosphate) | Arm B (Rituximab, Fludarabine Phosphate, Lenalidomide) | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide) | Arm D (Rituximab, Fludarabine, Cyclophosphamide, Lenalidomide)
Started | 138 | 140 | 140 | 0
Completed | 133 | 130 | 137 | 0
Not Completed | 5 | 10 | 3 | 0
Period: Re-assignment After Del(11q22.3) Testing
Arm/Group | Arm A (Rituximab, Fludarabine Phosphate) | Arm B (Rituximab, Fludarabine Phosphate, Lenalidomide) | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide) | Arm D (Rituximab, Fludarabine, Cyclophosphamide, Lenalidomide)
Started | 123 | 109 | 137 | 31
Completed | 123 | 109 | 137 | 31
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 400 participants were evaluable for analysis. (18 participants were excluded from the analysis.)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Rituximab, Fludarabine Phosphate) | Arm B (Rituximab, Fludarabine Phosphate, Lenalidomide) | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide) | Arm D (Rituximab, Fludarabine, Cyclophosphamide, Lenalidomide) | Total
Number analyzed (Participants) | 123 | 109 | 137 | 31 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 67 | 88 | 21 | 256
  >=65 years | 43 | 42 | 49 | 10 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 51 | 8 | 139
  Male | 83 | 69 | 86 | 23 | 261
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 14 | 16 | 8 | 53
  United States | 108 | 95 | 121 | 23 | 347

OUTCOME MEASURES:

1. Primary Outcome: 2-Year Progression Free Survival (PFS) Rate
Description: Proportion of participants who were alive and progression free at 2 years.
Time Frame: 2 years
Population: Patients re-assigned to Arm C were split into two analysis groups, patients with del(11q22.3), as assessed by interphase cytogenetics and present in at least 20% of cells, and those without del(11q22.3). This endpoint is limited to patients without del(11q22.3).
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Arm A, FR in Non-del(11q22.3): Participants, who are non-del(11q22.3), receive induction therapy (every 28 days for up to 6 cycles) of: rituximab (R) IV over 1-4 hours on days 1 (50 mg/m^2), 3 (325 mg/m^2), and 5 (375 mg/m^2) of course 1 and on day 1 (375 mg/m^2) of all subsequent courses. Patients also receive fludarabine phosphate (F) 25 mg/m^2/day IV over 30 minutes or PO on days 1-5.
- Arm B, FR+L in Non-del(11q22.3): Participants, who are non-del(11q22.3), receive induction therapy (every 28 days for up to 6 cycles) of: rituximab (R) IV over 1-4 hours on days 1 (50 mg/m^2), 3 (325 mg/m^2), and 5 (375 mg/m^2) of course 1 and on day 1 (375 mg/m^2) of all subsequent courses. Patients also receive fludarabine phosphate (F) 25 mg/m^2/day IV over 30 minutes or PO on days 1-5. Participants without progression receive consolidation therapy lenalidomide (L) 5mg/day cycle 1, 10 mg/day cycles 2-6 PO QD on days 1-21 of 28 day cycle.
- Arm C1, FCR in Non-del(11q22.3): Participants, who are non-del(11q22.3), receive induction therapy (every 28 days for up to 6 cycles) of: rituximab (R) IV over 4 hours on days 1 (50mg/m^2) and 3 (325 mg/m^2) of course 1 and on day 1 (500 mg/m^2) of all subsequent courses. Patients then receive fludarabine phosphate (F) (age < 70: 25 mg/m^2/day; age >= 70: 20 mg/m^2/day) IV piggyback over 30 minutes or PO (32 mg/m^2/day) followed by cyclophosphamide (C) (age < 70: 250 mg/m^2/day; age >= 70: 150 mg/m^2/day) IV piggyback over 30 minutes on days 1-3.
Arm/Group | Arm A, FR in Non-del(11q22.3) | Arm B, FR+L in Non-del(11q22.3) | Arm C1, FCR in Non-del(11q22.3)
Number analyzed (Participants) | 123 | 109 | 110
proportion of participants | 0.64 [0.57 to 0.71] | 0.71 [0.63 to 0.78] | 0.74 [0.66 to 0.80]

2. Secondary Outcome: Overall Response Rate in Patients Without Del(11q22.3)
Description: Percentage of non-del(11q22.3) participants with a complete response (CR) or partial response (PR). CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus >= 1 of the following: >= 1500/uL polymorphonuclear leukocytes, > 100,000/uL platelets, > 11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions.
Time Frame: Up to 15 years
Population: Patients without Del(11q22.3) were included in this analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Rituximab, Fludarabine Phosphate) | Arm B (Rituximab, Fludarabine Phosphate, Lenalidomide) | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide)
Number analyzed (Participants) | 123 | 109 | 110
percentage of participants | 75 [68 to 81] | 69 [61 to 76] | 71 [63 to 78]

3. Secondary Outcome: Overall Response Rates in Patients With Del(11q22.3)
Description: Percentage of del(11q22.3) participants with a complete response (CR) or partial response (PR). CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus >= 1 of the following: >= 1500/uL polymorphonuclear leukocytes, > 100,000/uL platelets, > 11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions.
Time Frame: Up to 15 years
Population: Patients with del(11q22.3) were included in this analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide) | Arm D (Rituximab, Fludarabine, Cyclophosphamide, Lenalidomide)
Number analyzed (Participants) | 27 | 31
percentage of participants | 59 [42 to 75] | 74 [58 to 86]

4. Secondary Outcome: PFS Rate of Patients With Del(11q22.3)
Description: Proportion of del (11q22.3) participants who were alive and progression free at 2 years.
Time Frame: 2 years
Population: This endpoint is limited to patients with del(11q22.3).
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Arm C2, FCR in Del(11q22.3): Participants who have del(11q22.3) receive induction therapy (every 28 days for up to 6 cycles) of: rituximab IV over 4 hours on days 1 (50mg/m^2) and 3 (325 mg/m^2) of course 1 and on day 1 (500 mg/m^2) of all subsequent courses. Patients then receive fludarabine phosphate (age < 70: 25 mg/m^2/day; age >= 70: 20 mg/m^2/day) IV piggyback over 30 minutes or PO (32 mg/m^2/day) followed by cyclophosphamide (age < 70: 250 mg/m^2/day; age >= 70: 150 mg/m^2/day) IV piggyback over 30 minutes on days 1-3.
- Arm D, FCR+L in Del(11q22.3): Patients who have del(11q22.3)receive the first course of induction therapy as in Arm A or B before being re-assigned to Arm D. Beginning in course 2, patients receive rituximab IV (500 mg/m^2) on day 1 and fludarabine phosphate (age < 70: 25 mg/m^2/day; age >= 70: 20 mg/m^2/day) IV piggyback over 30 minutes or PO (32 mg/m^2/day) and cyclophosphamide IV (age < 70: 250 mg/m^2/day; age >= 70: 150 mg/m^2/day) piggyback over 30 minutes on days 1-3. Participants without progression receive consolidation therapy: lenalidomide 5mg/day cycle 1, 10 mg/day cycles 2-6PO QD on days 1-21 of 28 day cycle.
Arm/Group | Arm C2, FCR in Del(11q22.3) | Arm D, FCR+L in Del(11q22.3)
Number analyzed (Participants) | 27 | 31
proportion of participants | 0.56 [0.38 to 0.72] | 0.65 [0.48 to 0.79]

5. Secondary Outcome: Time-to-progression in Patients Without Del(11q22.3)
Description: Time to progression (TTP) was defined as the registration date to date of progression or death due to any cause, whichever occurs first. TTP was estimated using the Kaplan Meier method. Progressive disease (PD) required at least one of the following: >= 50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes, >= 50% increase in the product of at least two lymphnodes, >= 50% increase in the enlargement of the liver and/or spleen.
Time Frame: Up to 15 years
Population: This endpoint is limited to patients without del(11q22.3).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A, FR in Non-del(11q22.3) | Arm B, FR+L in Non-del(11q22.3) | Arm C1, FCR in Non-del(11q22.3)
Number analyzed (Participants) | 123 | 109 | 110
months | 43.5 [32.8 to 49.9] | 66.0 [44.5 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment | 78.0 [57.9 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment

6. Secondary Outcome: Time-to-progression in Patients With Del(11q22.3)
Description: Time to progression (TTP) in del(11q22.3) participants was defined as the registration date to date of progression or death due to any cause, whichever occurs first. TTP was estimated using the Kaplan Meier method.
Time Frame: Up to 15 years
Population: This endpoint is limited to patients with del(11q22.3).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C2, FCR in Del(11q22.3) | Arm D, FCR+L in Del(11q22.3)
Number analyzed (Participants) | 27 | 31
months | 35.5 [21.8 to 65.5] | 44.6 [25.7 to 50.7]

ADVERSE EVENTS:
Arm/Group | Arm A (Rituximab, Fludarabine Phosphate) | Arm B (Rituximab, Fludarabine Phosphate, Lenalidomide) | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide) | Arm D (Rituximab, Fludarabine, Cyclophosphamide, Lenalidomide)
Serious Adverse Events (participants affected / at risk) | 13/123 | 21/109 | 14/137 | 3/31
Other Adverse Events (participants affected / at risk) | 117/123 | 107/109 | 132/137 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Rituximab, Fludarabine Phosphate) (N=123) | Arm B (Rituximab, Fludarabine Phosphate, Lenalidomide) (N=109) | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide) (N=137) | Arm D (Rituximab, Fludarabine, Cyclophosphamide, Lenalidomide) (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (6) | 4 (4) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (8) | 15 (17) | 10 (10) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 7 (7) | 2 (2) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (8) | 15 (17) | 6 (6) | 1 (1)
Fever (General disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (1) | 7 (7) | 5 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (7) | 12 (14) | 8 (8) | 0 (0)
Platelet count decreased (Investigations) | 9 (9) | 10 (12) | 9 (9) | 0 (0)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2) | 9 (9) | 4 (4) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Renal tubular disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 3 (3) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 2 (2) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Rituximab, Fludarabine Phosphate) (N=123) | Arm B (Rituximab, Fludarabine Phosphate, Lenalidomide) (N=109) | Arm C (Rituximab, Fludarabine Phosphate, Cyclophosphamide) (N=137) | Arm D (Rituximab, Fludarabine, Cyclophosphamide, Lenalidomide) (N=31)
Blood disorder (Blood and lymphatic system disorders) | 8 (22) | 5 (21) | 8 (26) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (17) | 13 (13) | 18 (18) | 5 (6)
Hemoglobin decreased (Blood and lymphatic system disorders) | 92 (398) | 90 (436) | 116 (516) | 23 (91)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 6 (16) | 0 (0) | 2 (4) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 4 (8) | 2 (6) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (5) | 9 (9) | 3 (4) | 2 (2)
Ventricular bigeminy (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 4 (5) | 3 (8) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 5 (16) | 0 (0) | 1 (6) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (3) | 0 (0) | 2 (4) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Eye pain (Eye disorders) | 3 (6) | 1 (2) | 1 (4) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flashing vision (Eye disorders) | 1 (1) | 2 (6) | 1 (2) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (4)
Retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 6 (7) | 8 (10) | 4 (4) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 4 (7) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 17 (22) | 18 (26) | 23 (24) | 4 (5)
Anal exam abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 35 (90) | 47 (123) | 46 (89) | 10 (23)
Diarrhea (Gastrointestinal disorders) | 30 (47) | 35 (88) | 39 (60) | 6 (15)
Dry mouth (Gastrointestinal disorders) | 4 (6) | 4 (10) | 1 (1) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (17) | 15 (24) | 10 (24) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 2 (9) | 1 (1) | 5 (6) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (2) | 6 (17) | 4 (5) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 3 (3) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (3) | 2 (2) | 3 (3) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (6) | 3 (3) | 3 (3) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 4 (15) | 3 (4) | 4 (8) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 8 (11) | 6 (10) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 64 (158) | 57 (155) | 79 (197) | 22 (50)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (9) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 3 (10) | 1 (1) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (5) | 3 (6) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 23 (41) | 17 (31) | 47 (74) | 5 (9)
Chest pain (General disorders) | 13 (14) | 13 (19) | 21 (30) | 1 (1)
Chills (General disorders) | 39 (50) | 39 (57) | 44 (61) | 5 (6)
Edema limbs (General disorders) | 15 (31) | 20 (41) | 20 (49) | 3 (10)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 89 (401) | 90 (481) | 106 (408) | 24 (119)
Fever (General disorders) | 19 (20) | 23 (27) | 23 (29) | 7 (8)
Flu-like symptoms (General disorders) | 0 (0) | 6 (10) | 4 (5) | 2 (2)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General symptom (General disorders) | 3 (3) | 1 (1) | 3 (6) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (4)
Localized edema (General disorders) | 3 (3) | 4 (4) | 10 (14) | 1 (2)
Pain (General disorders) | 12 (16) | 18 (38) | 19 (26) | 1 (1)
Pericardial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 2 (4) | 0 (0) | 2 (4) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 6 (6) | 5 (5) | 3 (3) | 1 (1)
Hypersensitivity (Immune system disorders) | 7 (7) | 11 (16) | 11 (13) | 2 (2)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 3 (3) | 2 (2) | 2 (3) | 1 (1)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 9 (11) | 11 (13) | 5 (7) | 1 (1)
Catheter related infection (Infections and infestations) | 3 (5) | 0 (0) | 4 (4) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Corneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 3 (4) | 1 (5) | 1 (1)
Eye infection intraocular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 7 (16) | 9 (12) | 4 (5) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 2 (3) | 4 (5) | 3 (3) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (5) | 2 (4) | 0 (0)
Opportunistic infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (10) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (10) | 8 (9) | 5 (5) | 2 (2)
Rhinitis infective (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 13 (18) | 12 (24) | 8 (11) | 0 (0)
Skin infection (Infections and infestations) | 8 (9) | 7 (10) | 8 (10) | 1 (1)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 15 (20) | 13 (21) | 12 (14) | 2 (3)
Ureteritis (Infections and infestations) | 10 (13) | 8 (9) | 9 (13) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (5) | 6 (8) | 9 (12) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Viral hepatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 6 (20) | 6 (6) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (7) | 1 (1) | 0 (0)
Intraoperative neurological injury - NERVES: Sciatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous injury - Extremity-upper (Injury, poisoning and procedural complications) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 3 (4) | 1 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 28 (74) | 29 (89) | 33 (89) | 7 (19)
Alkaline phosphatase increased (Investigations) | 19 (39) | 15 (42) | 23 (50) | 4 (4)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 31 (67) | 33 (76) | 33 (72) | 7 (13)
Blood bilirubin increased (Investigations) | 24 (59) | 17 (49) | 9 (9) | 4 (19)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 3 (3) | 4 (7) | 1 (6)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 22 (34) | 18 (34) | 19 (39) | 2 (3)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haptoglobin decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (4) | 2 (3) | 6 (18) | 0 (0)
Laboratory test abnormal (Investigations) | 8 (22) | 8 (20) | 11 (30) | 3 (3)
Leukocyte count decreased (Investigations) | 64 (258) | 61 (271) | 64 (273) | 14 (67)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 49 (225) | 48 (216) | 55 (281) | 10 (58)
Neutrophil count decreased (Investigations) | 100 (356) | 97 (420) | 109 (370) | 28 (106)
Platelet count decreased (Investigations) | 95 (528) | 85 (470) | 114 (546) | 22 (116)
Serum cholesterol increased (Investigations) | 2 (2) | 2 (5) | 2 (7) | 0 (0)
Weight gain (Investigations) | 13 (31) | 13 (21) | 12 (29) | 1 (1)
Weight loss (Investigations) | 5 (5) | 12 (15) | 10 (16) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 23 (41) | 28 (49) | 20 (26) | 7 (16)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (6) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 54 (185) | 54 (217) | 62 (212) | 10 (39)
Blood uric acid increased (Metabolism and nutrition disorders) | 7 (12) | 9 (22) | 10 (16) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 2 (6) | 2 (2) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (11) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 15 (23) | 23 (43) | 20 (29) | 4 (12)
Serum calcium decreased (Metabolism and nutrition disorders) | 31 (59) | 42 (78) | 38 (68) | 7 (20)
Serum calcium increased (Metabolism and nutrition disorders) | 4 (7) | 5 (10) | 2 (8) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 6 (14) | 5 (12) | 8 (10) | 1 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 3 (5) | 6 (14) | 6 (7) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 12 (23) | 15 (36) | 8 (13) | 3 (5)
Serum potassium decreased (Metabolism and nutrition disorders) | 16 (33) | 19 (35) | 22 (36) | 3 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 11 (13) | 10 (14) | 12 (15) | 1 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 21 (40) | 28 (46) | 23 (44) | 3 (3)
Serum sodium increased (Metabolism and nutrition disorders) | 7 (8) | 1 (1) | 2 (5) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (65) | 24 (57) | 24 (53) | 3 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (4) | 6 (13) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (28) | 21 (57) | 23 (44) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (11) | 7 (8) | 7 (11) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 4 (6) | 1 (1)
Fibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 3 (11) | 2 (3) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (11) | 10 (12) | 3 (10) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (11) | 1 (2) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 5 (7) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (31) | 15 (43) | 16 (25) | 4 (5)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 5 (8) | 11 (20) | 2 (2)
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (34) | 18 (39) | 16 (33) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 8 (16) | 5 (8) | 0 (0)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (5)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 17 (33) | 25 (49) | 19 (32) | 2 (5)
Dysgeusia (Nervous system disorders) | 9 (14) | 12 (19) | 5 (6) | 1 (4)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 2 (3) | 3 (3) | 1 (2)
Headache (Nervous system disorders) | 33 (62) | 35 (72) | 27 (60) | 8 (22)
Memory impairment (Nervous system disorders) | 3 (3) | 3 (22) | 5 (9) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 4 (6) | 5 (10) | 7 (12) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (39) | 20 (69) | 17 (56) | 2 (3)
Phrenic nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 4 (4) | 3 (6) | 2 (2) | 0 (0)
Speech disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (4) | 3 (4) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 3 (10) | 3 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 14 (38) | 17 (27) | 13 (22) | 2 (4)
Confusion (Psychiatric disorders) | 1 (2) | 2 (3) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 8 (35) | 11 (23) | 9 (16) | 2 (18)
Euphoria (Psychiatric disorders) | 0 (0) | 2 (8) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 19 (45) | 23 (52) | 25 (55) | 5 (12)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (6) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 2 (5) | 3 (3) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (7) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 5 (10) | 2 (2) | 0 (0)
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 6 (7) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 6 (15) | 9 (17) | 12 (21) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 3 (3) | 4 (16) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 5 (9) | 4 (10) | 5 (15) | 2 (3)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (7) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 18 (48) | 18 (42) | 13 (24) | 1 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (7) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (69) | 48 (122) | 44 (91) | 8 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 32 (102) | 43 (104) | 43 (90) | 9 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (8) | 4 (7) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (6) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (2) | 2 (2) | 0 (0)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (14) | 8 (19) | 13 (16) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (10) | 1 (4) | 2 (4)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (9) | 4 (16) | 3 (5) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 10 (21) | 6 (21) | 2 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (5) | 2 (3) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (24) | 20 (35) | 18 (25) | 7 (14)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 32 (48) | 49 (122) | 50 (99) | 15 (28)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (11) | 9 (14) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 21 (52) | 27 (50) | 31 (81) | 6 (12)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (9) | 4 (7) | 6 (8) | 1 (1)
Flushing (Vascular disorders) | 4 (9) | 7 (17) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 4 (9) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 5 (9) | 3 (10) | 6 (14) | 2 (6)
Hypertension (Vascular disorders) | 16 (27) | 18 (76) | 20 (55) | 1 (1)
Hypotension (Vascular disorders) | 15 (24) | 12 (13) | 20 (30) | 2 (2)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Phlebitis (Vascular disorders) | 5 (6) | 1 (3) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less